CLINICAL TRIAL: NCT04953390
Title: Evaluating Benefits of Hearing Aid Microphone Directionality Technologies on Spatial Awareness and Speech Intelligibility
Brief Title: Evaluating Benefits of Hearing Aid Microphone Directionality Technologies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SRF-369
Record Dates: First submitted 2021-06-09; First posted 2021-07-08 (Actual); Results first posted 2022-11-09 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2021-07

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Intervention Model Description: A single group of participants will be evaluating different directional microphone settings on commercially available hearing aids
Masking Description: During lab testing, participants will be aware of the device they are wearing, but will not be aware of which microphone setting is being tested.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Experimental (Experimental): All study participants wearing study devices and evaluating three different microphone settings in simulated noise environments in lab, and using study devices during home trial period.
  Interventions: Device: Phonak Audeo hearing aid; Device: Phonak hearing aid with multiple directionality settings, adjustable via a mobile app

INTERVENTIONS:
Device: Phonak Audeo hearing aid — Commercially available hearing aid with three different microphone settings: DIR1, DIR2, and DIR3
Device: Phonak hearing aid with multiple directionality settings, adjustable via a mobile app — Commercially available hearing aid with multiple directionality settings which will be adjustable by user via a mobile app during a home trial period.

SUMMARY:
This study will evaluate the impact of hearing aid microphone directionality technologies and settings on speech understanding in noise for experienced hearing aid users. It will also evaluate the participant's spatial awareness of sounds using these different hearing aid microphone directionality technologies.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* experienced hearing aid users
* moderate to moderate severe sensorineural symmetrical hearing loss defined as a difference of less than 10 dB between ears
* must be able to use app and smart phone

Exclusion Criteria:

* asymmetrical hearing losses
* unable or unwilling to use app and smart phone

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2021-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Seitz-Paquette, AuD, Principal Investigator — Sonova AG
Locations (1):
- Sonova, Aurora, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants who were tested using different microphone directionality settings.
Arm/Group | Experimental
Number analyzed (Participants) | 19
Age, Continuous [Mean (Full Range); unit: years] | 72 [39 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 19
Hearing Loss [Count of Participants; unit: Participants] — All participants with a moderate to moderately severe sensorineural hearing loss, as measured by a recent (less than 12 months) audiogram.
  Participants | 19

OUTCOME MEASURES:

1. Primary Outcome: Subjective Description of DIR1, DIR2, and DIR3 in Controlled Soft Noise Environment
Description: Participant describes an acoustically noisy environment in which recorded speech is played from a speaker directly in front of the participant and recorded multi-talker babble is played from multiple speakers around the participant. The participant uses a slider tool to choose if scene sounds acoustically wide (hearing all noise and speech), or acoustically narrow (hearing more of the speech than the noise). The range of the slider is 0-100, with 0 indicating the sound scene is "wide" and 100 indicating the sound scene is "narrow". The slider moves in 5 point increments. This is a purely subjective description and there is no better or worse outcome.
Time Frame: Third appointment (day 28 of study)
Population: Participants who were able to complete the tasks as instructed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental
Number analyzed (Participants) | 16
units on a scale
  Perceived narrowness of DIR1 in soft noise | 40.31 (24.73)
  Perceived narrowness DIR2 in soft noise | 55.94 (19.99)
  Perceived narrowness DIR3 in soft noise | 66.88 (18.81)
Statistical Analysis 1: Comparison: Experimental; Test type: Other; p = 0.004, ANOVA

2. Primary Outcome: Subjective Description of DIR1, DIR2, and DIR3 in Controlled Loud Noise Environment
Description: as for outcome 1
Time Frame: Third appointment (day 28 of study)
Population: Participants who were able to complete the task
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental
Number analyzed (Participants) | 16
units on a scale
  Perceived narrowness DIR1 in loud noise | 35.31 (26.23)
  Perceived narrowness DIR2 in loud noise | 48.91 (22.71)
  Perceived narrowness DIR3 in loud noise | 57.5 (19.26)
Statistical Analysis 1: Comparison: Experimental; Test type: Other; p = .029, ANOVA

3. Primary Outcome: Subjective Preference DIR1, DIR2, and DIR3 in Controlled Soft Noise Environments
Description: Using a sliding scale, the participant chooses their preference for listening to the sound scene, however this time, 0 indicates "not preferred" and 100 indicates "most preferred". The slider moves in 5 point increments. This is purely subjective and there is no better or worse answer.
Time Frame: Third appointment (day 28 of study)
Population: All study participants who were able to complete task.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental
Number analyzed (Participants) | 16
units on a scale
  Preference for DIR1 in soft noise | 31.41 (24.22)
  Preference for DIR2 in soft noise | 53.13 (21.03)
  Preference for DIR3 in soft noise | 64.1 (16.28)
Statistical Analysis 1: Comparison: Experimental; Test type: Other; p = 0.0002, ANOVA

4. Secondary Outcome: Speech Reception Threshold
Description: Objective measure of speech reception thresholds with all three microphone settings (DIR1,DIR2,DIR3). This is calculated as the Signal to Noise Ratio at which participant can correctly repeat 50% of the words. A negative number (i.e. -10) indicates that the participant correctly repeated 50% of the words when the speech signal was softer or lower than the noise level. For example, an SNR score of -10 means that the the participant correctly repeated 50% of the words when the speech signal was 10 dB softer than the noise level. In this case, the noise level was appropriate to the microphone setting, i.e., DIR1 was tested in softer noise and DIR2 and DIR3 were tested in loud noise.
Time Frame: 2nd appointment (Day 14 of study)
Population: All participants who were able to complete the tasks as instructed.
Measure: Mean (Standard Deviation); unit: dB SNR
Arm/Group | Experimental
Number analyzed (Participants) | 17
dB SNR
  SNR level for DIR1 in soft noise | -10.22 (2.4)
  SNR level for DIR2 in loud noise | -12.35 (1.75)
  SNR level for DIR3 in loud noise | -11.85 (1.94)
Statistical Analysis 1: Comparison: Experimental; All three DIR settings were tested, but only the DIR2 and DIR3 were compared in t-test. This is because DIR1 mic setting was tested in a different condition (i.e. softer noise); Test type: Other; p = .14, t-test, 2 sided; T-test done on DIR2 and DIR3 results only, as the conditions were equal for these two settings. DIR1 was tested in a different condition

5. Secondary Outcome: Observations and Ratings of Satisfaction of Microphone Directionality in Real Life
Description: Participants made adjustments of microphone directionality via an app, in real world listening situations. When participants adjusted the microphone directionality in real-time, they were also prompted via ecological momentary assessment to rate how satisfied they were with the adjustment. Participants chose one of three satisfaction ratings: no, slight, or clear. "Clear" satisfaction would be the best rating, indicating high satisfaction, "no" would be the worst rating, indicating no satisfaction, and "slight" would indicate somewhat satisfied.
Time Frame: 4 weeks
Population: All participants who wore devices in real world situations during a four week time period, and who were able to access and operate the mobile app.
Measure: Number; unit: adjustments
Units Other Than Participants: adjustments
Arm/Group | Experimental
Number analyzed (Participants) | 19
Number analyzed (adjustments) | 255
adjustments
  Number of adjustments in which user rated "clear" satisfaction | 113
  Number of adjustments in which users rated "slight" satisfaction | 95
  Number of adjustments in which user rated "no" satisfaction | 47

6. Secondary Outcome: Subjective Ratings of Transition Speed From One Directional Microphone Setting to Another Directional Setting
Description: Participants listen to different samples of transition speed from one mic setting to another in an A/B comparison and rate which sample is more noticeable, i.e. A is more noticeable than B, A is less noticeable than B, or A and B are the same. No statistical analysis was done for this outcome measure. Frequency distribution was completed to record the number of responses in which participants rated a 0 second transition time more noticeable than a 2s, 4s, and 8s transition time.
Time Frame: Third appointment (day 28 of study)
Population: All participants who were able to complete the task as instructed.
Measure: Number; unit: comparisons between two time constants
Units Other Than Participants: responses
Arm/Group | Experimental
Number analyzed (Participants) | 19
Number analyzed (responses) | 114
comparisons between two time constants
  Number of times 0 seconds is rated as more noticeable than 2,4,or 8 seconds | 58
  Number of times 0 seconds is rated as no different than 2,4, or 8 seconds | 29
  Number of times 0 seconds is rated as less noticeable than 2,4, or 8 seconds | 27

7. Primary Outcome: Subjective Preference DIR1, DIR2, and DIR3 in Controlled Loud Noise Environments
Description: Using a sliding scale, the participant chooses their preference for listening to the sound scene, however this time, 0 indicates "not preferred" and 100 indicates "most preferred". The slider moves in 5 point increments.
Time Frame: Third appointment (day 28 of study)
Population: All study participants who were able to complete task as instructed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental
Number analyzed (Participants) | 16
units on a scale
  Preference for DIR1 in loud noise | 26.25 (26)
  Preference for DIR2 in loud noise | 43.75 (20.43)
  Preference for DIR3 in loud noise | 60.78 (19.81)
Statistical Analysis 1: Comparison: Experimental; Test type: Other; p = .0003, ANOVA

ADVERSE EVENTS:
Time Frame: 4-6 weeks
Arm/Group | Experimental
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-24): https://cdn.clinicaltrials.gov/large-docs/90/NCT04953390/Prot_SAP_000.pdf